CLINICAL TRIAL: NCT04469075
Title: The PROTECT Study: A Phase II, Open-Label Trial of PROphylactic Skin Toxicity ThErapy With Clindamycin and Triamcinolone in Glioblastoma Patients Treated With Tumor Treating Fields
Brief Title: Clindamycin and Triamcinolone in People With Glioblastoma to Prevent Skin-Related Side Effects of Tumor Treating Fields
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-342
Record Dates: First submitted 2020-07-10; First posted 2020-07-13 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; Skin Toxicity
Keywords: Clindamycin; Triamcinolone; Skin-Related Side Effects; Recurrent; 19-342
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — clindamycin phosphate; Triamcinolone Acetonide

STUDY DESIGN:
Intervention Model Description: This is a phase 2, multicenter, open-label study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- topical clindamycin and triamcinolone (Experimental): Patients who are scheduled to receive TTFields therapy for newly diagnosed GBM will be treated with: topical clindamycin (or approved equivalent) 1% and triamcinolone 0.1%. Participating sites may use an alternative equivalent form of clindamycin, such as a gel, with MSK PI approval
  Interventions: Drug: Clindamycin Phosphate; Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Clindamycin Phosphate — phosphate 1% solution triamcinolone 0.01% at every array change (or approved equivalent)
Drug: Triamcinolone Acetonide — triamcinolone acetonide 0.01% lotion triamcinolone 0.01% at every array change

SUMMARY:
The participants are being treated with Tumor Treating Fields (TTFields) for malignant glioma, and this type of treatment may cause skin-related side effects. This study will test whether using clindamycin and triamcinolone topical lotions can prevent skin-related side effects of TTFields.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of newly diagnosed or recurrent GBM with plan to initiate treatment with TTFields with or without systemic therapy, confirmed by the enrolling institution
* Able to self-administer topical interventions or has available another person who can apply the topical agents
* Treatment with TTF should be initiated within 7 days of planned initiation on this trial.

Exclusion Criteria:

* Known history of allergy to any ingredient of the study agents
* Preexisting scalp disorders such as psoriasis or dermatitis that, in the opinion of the investigator, will affect the grading of skin adverse events, confirmed by enrolling institution.
* Use of concurrent topical therapy to the scalp for another dermatologic condition
* Active, uncontrolled infection requiring systemic or oral antibiotic therapy within 14 days of enrollment
* Use of greater than 4 mg dexamethasone a day within 14 days of enrollment
* Malignant glioma
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients without grade 2 or higher skin toxicity | up to 120 days
  device-related skin adverse events by investigator assessment.

SECONDARY OUTCOMES:
skin-related quality of life | up to 120 days
  using the PRO-CTCAE for rash, ulcer, and pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Northwestern University, Evanston, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center Suffolk - Hauppauge (All Protocol Activities), Hauppauge, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm